CLINICAL TRIAL: NCT02791490
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Study the Safety and Efficacy of the Addition of Sitagliptin During Metformin Up-titration Compared With Metformin Up-titration Alone in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study of the Safety and Efficacy of Sitagliptin Addition During Metformin Up-titration (MK-0431-848)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-848; MK-0431-848 (Other: Merck); 2015-004224-59 (EudraCT Number)
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Sitagliptin (Experimental): Participants will receive sitagliptin 100 mg once daily for 20 weeks. They will also receive immediate-release metformin (Met-IR), which will be titrated from a baseline dose of 1000 mg/day (500 mg/twice a day [b.i.d.]) up to 2000 mg/day (1000 mg/b.i.d.) by Day 15. Participants will also receive glycemic rescue therapy as needed.
  Interventions: Drug: Sitagliptin; Drug: Metformin IR
- Placebo (Placebo Comparator): Participants will receive placebo matching sitagliptin once daily for 20 weeks. They will also receive Met-IR, which will be titrated from baseline dose of 1000 mg/day (500 mg/b.i.d.) up to 2000 mg/day (1000 mg/b.i.d.) by Day 15. Participants will also receive glycemic rescue therapy as needed.
  Interventions: Drug: Placebo; Drug: Metformin IR

INTERVENTIONS:
Drug: Sitagliptin — Oral tablet, 100 mg, once daily at approximately the same time each day
  Other Names: JANUVIA®; TESAVEL®; XELEVIA®; RISTABEN®
  Arms: Sitagliptin
Drug: Placebo — Oral tablet, once daily at approximately the same time each day
  Arms: Placebo
Drug: Metformin IR — All participants will take Met-IR as background medication. Initially, they will take 1 x 500 mg tablet Met-IR b.i.d. (1000 mg/day). After randomization, all participants will be titrated to 2 x 500 mg tablets of Met-IR b.i.d. (2000 mg/day).

SUMMARY:
This trial is designed to evaluate, in adult participants with Type 2 diabetes mellitus (T2DM) and inadequate glycemic control on sub-maximal metformin mono-therapy (1000 mg/day), the effect of up-titration of metformin plus the addition of sitagliptin compared to up-titration of metformin alone on glycemic control. The primary hypothesis of this study is that up-titration of metformin to 2000 mg/day (1000 mg/twice a day) plus the addition of sitagliptin 100 mg/day provides greater reduction in hemoglobin A1C (A1C) compared to metformin up-titration alone. Another primary objective of this study is to evaluate the safety and tolerability of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants with T2DM in accordance with American Diabetes Association (ADA) guidelines
* Meet one of the following criteria:

  1. Be on stable Met-IR monotherapy 1000 mg/day for ≥8 weeks with a Screening A1C ≥7.5% and ≤11.0%.

     OR
  2. Be on stable Met-XR monotherapy 1000 mg/day for ≥8 weeks with a Screening A1C ≥7.5% and ≤11.0%.

     OR
  3. Not on any anti-hyperglycemic agent (AHA) for ≥8 weeks (≥12 weeks if previously taking thiazolidinediones) with a Screening A1C ≥8.5% and ≤12.0%.

     OR
  4. Be on stable monotherapy with a sulfonylurea, a glinide, or an α-glucosidase inhibitor for ≥8 weeks with a Screening A1C ≥7.5% and ≤11.0%.
* A body mass index (BMI) ≥18.0 kg/m2.
* Is a male or a female not of reproductive potential (defined as one who is postmenopausal or has had a hysterectomy and/or bilateral oophorectomy, or had bilateral tubal ligation or occlusion at least 6 weeks prior to Screening visit). If participant is a female of reproductive potential, must agree to remain abstinent from heterosexual activity or agrees to use (or have her partner use) acceptable contraception to prevent pregnancy while receiving blinded study drug and for 14 days after the last dose of blinded study drug

Exclusion Criteria:

* Has a history of type 1 diabetes mellitus or a history of ketoacidosis or has a history of secondary causes of diabetes (e.g., genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrinopathies, drug- or chemical-induced, and post-organ transplant).
* A known hypersensitivity or intolerance to any DPP-4 inhibitor. A known hypersensitivity or intolerance to metformin, including participants who were previously unable to tolerate metformin at a dose >1000 mg/day or who have evidence of intolerance to the dose of metformin they are currently taking.
* Has been treated with any of the following agents within 8 weeks (12 weeks for thiazolidinediones) of study participation:

  1. Insulin of any type (except for short-term use [i.e., ≤7 days] during concomitant illness or other stress)
  2. DPP-4 inhibitor
  3. Pioglitazone or rosiglitazone (thiazolidinediones)
  4. Glucagon-like peptide-1 receptor (GLP-1R) agonists
  5. Sodium glucose co-transporter 2 (SGLT2) inhibitors
  6. Bromocriptine (Cycloset™)
  7. Colesevelam (Welchol™)
  8. Any other AHA with the exception of protocol-approved agents
* Intends to initiate weight loss medication during the study period
* Has undergone bariatric surgery within 12 months of Screening visit
* Has started a weight loss medication or a medication associated with weight changes within the prior 12 weeks
* A history of myocardial infarction, unstable angina, arterial revascularization, stroke, transient ischemic attack, NYHA functional class III-IV heart failure, or severe peripheral vascular disease (e.g., claudication with minimal activity, a nonhealing ischemic ulcer, or disease which is likely to require surgery or angioplasty) within 3 months of study participation
* A history of malignancy ≤5 years prior to study participation (i.e., the diagnosis occurred, or any evidence of residual or recurrent disease occurred, within the past 5 years), except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer. Note: A patient with any history of melanoma, leukemia, lymphoma, or renal cell carcinoma is excluded.
* Has human immunodeficiency virus (HIV)

  1. with AIDS related complications, or
  2. has not been on a stable anti-retroviral regimen for >6 months, or
  3. has progressive disease, or
  4. using agents associated with glucose intolerance such as nucleoside reverse transcriptase inhibitors (NRTIs) such as azidothymidine (AZT), didanosine (ddI), and stavudine (d4T).
* Is on or likely to require treatment for ≥14 consecutive days or repeated courses of pharmacologic doses of corticosteroids.
* Has undergone a major surgical procedure within 12 weeks prior to signing the informed consent form (ICF) or has major surgery planned during the trial.
* Currently participating, or has participated, in a study in which the participant received an investigational compound or used an investigational device within the prior 12 weeks of signing informed consent or is not willing to refrain from participating in another study.
* Is pregnant or breast-feeding, has a positive urine pregnancy test, or is planning to conceive or donate eggs during the study, including 14 days following the last dose of blinded investigational product.
* A recent history of alcohol or drug abuse (within 3 years) or is a user of recreational or illicit drugs at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Frias JP, Zimmer Z, Lam RLH, Amorin G, Ntabadde C, Iredale C, O'Neill EA, Engel SS, Kaufman KD, Makimura H, Crutchlow MF. Double-blind, randomized clinical trial assessing the efficacy and safety of early initiation of sitagliptin during metformin uptitration in the treatment of patients with type 2 diabetes: The CompoSIT-M study. Diabetes Obes Metab. 2019 May;21(5):1128-1135. doi: 10.1111/dom.13626. Epub 2019 Feb 17. PMID 30609212

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin: Participants received sitagliptin 100 mg once daily for 20 weeks. They also received immediate-release metformin (Met-IR), which was titrated from a baseline dose of 1000 mg/day (500 mg/twice a day [b.i.d]) up to 2000 mg/day (1000 mg/b.i.d.) by Day 15. Participants also received glycemic rescue therapy as needed.
- Placebo: Participants received placebo matching sitagliptin once daily for 20 weeks. They also received Met-IR, which was titrated from baseline dose of 1000 mg/day (500 mg/b.i.d.) up to 2000 mg/day (1000 mg/b.i.d.) by Day 15. Participants also received glycemic rescue therapy as needed.
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 229 | 229
Completed | 226 | 221
Not Completed | 3 | 8
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Sitagliptin: Participants received sitagliptin 100 mg once daily for 20 weeks. They also received Met-IR, which was titrated from a baseline dose of 1000 mg/day (500 mg/b.i.d.) up to 2000 mg/day (1000 mg/b.i.d.) by Day 15. Participants also received glycemic rescue therapy as needed.
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 229 | 229 | 458
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.6 (10.5) | 55.3 (10.4) | 55.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 136 | 275
  Male | 90 | 93 | 183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 147 | 151 | 298
  Not Hispanic or Latino | 78 | 70 | 148
  Unknown or Not Reported | 4 | 8 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 23 | 27 | 50
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 7 | 15
  White | 167 | 155 | 322
  More than one race | 31 | 39 | 70
  Unknown or Not Reported | 0 | 0 | 0
Hemoglobin A1C (%) [Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin] | 8.6 (0.9) | 8.7 (1.0) | 8.7 (0.9)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 181.7 (41.6) | 184.4 (44.7) | 183.0 (43.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C at Week 20
Description: Hemoglobin A1C is a blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. The change from baseline represents the Week 20 A1C value minus the Week 0 (baseline) A1C value.
Time Frame: Baseline and Week 20
Population: All randomized participants who received at least 1 dose of study medication and had at least 1 observation for the analysis endpoint
Measure: Least Squares Mean (95% Confidence Interval); unit: A1C (%)
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 229 | 229
A1C (%) | -1.10 [-1.28 to -0.93] | -0.69 [-0.88 to -0.51]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority; p < 0.001, Longitudinal Data Analysis; Difference in Least Squares Means = -0.41, 95% CI 2-sided [-0.59 to -0.23]

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event (AE)
Description: An adverse event (AE) is any untoward medical occurrence in a study participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to 22 weeks
Population: All randomized participants who received at least 1 dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 229 | 229
Percentage of participants | 44.1 | 45.9
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Other — 95% CI; Miettinen and Nurminen method; Difference in % vs Placebo = -1.7, 95% CI 2-sided [-10.8 to 7.4]

3. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: as for outcome 2
Time Frame: Up to 20 weeks
Population: All randomized participants who received at least 1 dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 229 | 229
Percentage of participants | 0.9 | 0.0

4. Secondary Outcome: Percentage of Participants With Hemoglobin A1C <7% at Week 20
Description: Hemoglobin A1C is a blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100.
Time Frame: Week 20
Population: All randomized participants who received at least 1 dose of study treatment and had at least 1 observation for the analysis endpoint
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 229 | 229
Percentage of participants | 28.8 | 16.6
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority; p = 0.002, Miettinen and Nurminen method; Relative Risk = 1.7, 95% CI 2-sided [1.2 to 2.5]

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 20
Description: Plasma glucose was measured on a fasting basis and is expressed as mg/dL. Blood was drawn predose on Day 1 and after 20 weeks of treatment to determine change in FPG levels. The change from baseline represents the Week 20 FPG value minus the Week 0 (baseline) FPG value.
Time Frame: Baseline and Week 20
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 229 | 229
mg/dL | -29.3 [-37.5 to -21.1] | -16.9 [-25.2 to -8.6]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority; p = 0.002, Longitudinal Data Analysis; Difference in Least Squares Means = -12.4, 95% CI 2-sided [-20.2 to -4.6]

6. Secondary Outcome: Percentage of Participants With Hemoglobin A1C ≥8.5% at Baseline That Attained A1C Goal of <7% at Week 20
Description: as for outcome 4
Time Frame: Baseline and Week 20
Population: The subgroup of randomized participants who had a baseline hemoglobin A1C ≥8.5%, received at least 1 dose of study medication, and had at least 1 observation for the analysis endpoint
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 122 | 122
Percentage of participants | 15.6 | 5.7

7. Secondary Outcome: Percentage of Participants Receiving Glycemic Rescue Therapy
Description: Participants who met pre-specified criteria for glycemic rescue received appropriate rescue therapy. The choice of anti-hyperglycemic rescue agent, dose, and regimen was directed by the investigator, as clinically appropriate.
Time Frame: Up to 20 weeks
Population: All randomized participants who received at least 1 dose of study treatment
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 229 | 229
Percentage of participants | 1.3 | 3.1

ADVERSE EVENTS:
Time Frame: Up to 22 weeks
Description: All randomized participants who received at least 1 dose of study medication
Arm/Group | Sitagliptin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/229 | 0/229
Serious Adverse Events (participants affected / at risk) | 3/229 | 4/229
Other Adverse Events (participants affected / at risk) | 18/229 | 11/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=229) | Placebo (N=229)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Fatty liver alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=229) | Placebo (N=229)
Diarrhoea (Gastrointestinal disorders) | 18 (18) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT02791490/Prot_SAP_000.pdf